CLINICAL TRIAL: NCT04874675
Title: A Randomised Control Clinical Trial Comparing Diclofenac / Acetaminophen /Codeine and Ibuprofen/Acetaminophen/Codeine Combination for Pain Management After Third Molars Surgery
Brief Title: An Randomized Control Trial Comparing Two Drug Combinations for Pain Management After Third Molars Surgery
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Covid 19 lockdown
Sponsor: University of Zimbabwe (Other)
Collaborators: UZ-CHS-PERFECT (Unknown)
Responsible Party: Principal Investigator, Silas Bere, Lecturer, University of Zimbabwe
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UZCHS PERFECT THIRD MOLAR
Record Dates: First submitted 2021-04-28; First posted 2021-05-06 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: Impacted Third Molar Tooth; PAIN
MeSH Terms: conditions — Pain | interventions — Diclofenac; Acetaminophen; Codeine; Ibuprofen; acetaminophen, codeine drug combination

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Diclofenac /Acetaminophen/Codeine (Active Comparator): routine pain medication used in post extraction pain management
  Interventions: Drug: diclofenac / acetaminophen /codeine
- Ibuprofen/Acetaminophen/codeine (Active Comparator): routine pain medication used in post extraction pain management
  Interventions: Drug: ibuprofen/acetaminophen/codeine

INTERVENTIONS:
Drug: diclofenac / acetaminophen /codeine — routine pain medication used post extraction of third molars
  Other Names: diclofenac/paracetamol/codeine phosphate
  Arms: Diclofenac /Acetaminophen/Codeine
Drug: ibuprofen/acetaminophen/codeine — routine pain medication used post extraction of third molars
  Other Names: ibuprofen/paracetamol/codeine phosphate
  Arms: Ibuprofen/Acetaminophen/codeine

SUMMARY:
Randomised control clinical trial to compare which combination of analgesics in effective in pain management after third molar extraction of wisdom teeth. The study will assess post operative pain after third molar extraction of two groups of study participants who will be given one of the two combinations of Diclofenac/ acetaminophen/codeine and ibuprofen/acetaminophen/codeine .

DETAILED DESCRIPTION:
Double blind randomized control clinical trial to compare the level of pain relief that occurs after third molar extraction done under local anaesthesia at the maxillofacial center, Harare, Zimbabwe. The participants will be randomized into two arms upon fitting the inclusion criteria.The pharmacist will be in charge of randomization and will randomise the participants upon giving them the medications. One group will receive combination of diclofenac/acetaminophen/codeine and the other group will receive ibuprofen/acetaminophen/codeine as post extraction analgesia.The dosages of the medications will be Diclofenac 50mg, ibuprofen 400mg, acetaminophen 500mg and codeine 15mg respectively. Questionnaires will be given to the patient to complete after discharge from the surgery and other parts of the questionnaire will be completed on review after 7 days. A record will be done of the postoperative pain experience (using visual analogue scale), use of rescue medication and details pertaining to impacted tooth.

ELIGIBILITY:
Inclusion Criteria:

* patients older than 18 years of age
* patients undergoing third molar extractions
* patients with or willing to get orthopantomogram for assessment of impacted third molars

Exclusion Criteria:

* patients younger than 18 years
* patients not willing to consent to the study
* patients with associated co-morbidities
* patients not willing to undergo radiological evaluation
* patients allergic to medications used in the study
* pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2023-03 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
post operative pain | within 7 days post extraction
  record of pain felt by patients on Visual analogue scale using a smiling face to show no pain and worst pain ever with a sad face measured line at 100mm . a score of 100mm indication worst pain and score of 0mm indicating no pain.

SECONDARY OUTCOMES:
Time rescue medication is used | within 7 days post extraction
  rescue medication
cheek swelling | with in 7 days post extraction
  amount of cheek swelling post extraction

CONTACTS AND LOCATIONS:
Locations (1):
- Dr Silas bere, Harare, Zimbabwe

IPD SHARING:
Plan to Share IPD: Undecided